CLINICAL TRIAL: NCT03795688
Title: The Role of Sex Steroids and Serotonin Brain Dynamics in Perinatal Mental Health
Status: Completed | Type: Observational
Sponsor: Vibe G Frøkjær, MD, PhD (Other)
Collaborators: Center for Integrated Molecular Brain Imaging, Copenhagen, Denmak (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Vibe G Frøkjær, MD, PhD, Senior researcher, Principal investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: PND1; H-18029563 (Other: Regional ethics committee)
Record Dates: First submitted 2018-12-18; First posted 2019-01-08 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Major Depressive Disorder; Perinatal Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Basic, non-imaging group: Pregnant women who will deliver by planned caesarian. Participants enrolled in the study that are not eligible for the imaging subgroup.
  All participants start in the basic program. Includes collection of blood, cerebrospinal fluid, saliva, hair, placenta tissues, umbilical cord blood and psychometrics.
  Interventions: Other: Pregnancy
- Extended, imaging group: A subgroup of 70 pregnant women who will deliver by planned caesarian selected towards either high (N=35) or low (N=35) risk for perinatal depression will undergo brain imaging in addition to the elements of the basic program. The extended imaging program includes functional and structural magnetic resonance imaging, positron emission tomography (PET) and a semistructured interview for depression symptoms (HAM-D17).
  Interventions: Other: Pregnancy

INTERVENTIONS:
Other: Pregnancy — Peripartum transition from pregnant to postpartum state

SUMMARY:
Hormonal transitions such as across pregnancy and postpartum may trigger depressive episodes in some women. It is not known why, but estrogen sensitivity may play a critical role. A preclinical human risk model showed that depressive symptoms induced by pharmacological sex-hormone manipulation is linked to increases in serotonin transporter (SERT) brain binding, which lowers serotonergic brain tone. It is currently unknown if these findings translates to women across pre- to postpartum transitions.

This longitudinal project studies a group of women who will deliver by planned caesarian, thus permitting the collection of cerebrospinal fluid (csf) containing central markers of serotonergic signaling, at the latest point in pregnancy. The women are followed across late pregnancy, delivery and 6 months postpartum to illuminate relations between sex-hormones, stress-regulation, estradiol sensitivity, csf markers of neurotransmission, serotonin transporter genotype variance, and potential development of subclinical or manifest depressive symptoms. Further, markers of relevance for the infant brain development and stress-regulation will be obtained from placenta tissue and umbilical cord blood. A subgroup of 70 women will participate in a brain imaging program early postpartum (week 3-5), which includes an evaluation of brain activity and structure and in vivo molecular brain imaging serotonergic markers. Thus, serotonergic markers in csf can be combined with postpartum molecular brain imaging of key features of serotonin signaling. Women in the imaging program are selected based on variation in their level of mental distress immediately postpartum (day 2-5).

The study's main hypothesis is that women with high-expressing SERT genotypes are more sensitive to peripartum hormonal transition in terms of changes in serotonergic tone and emergence of depressive symptoms and that such an association will be stronger in the presence of candidate gene transcript biomarkers of oestrogen sensitivity. A further hypothesis is that in vivo molecular brain imaging and csf based serotonergic markers will be associated with depressive symptoms both early and later postpartum.

Ideally, this project will provide a rationale for future targeted prevention and/or treatment of perinatal depression in women at high risk, which holds grand potential to protect not only mother but also infant brain health long-term.

DETAILED DESCRIPTION:
Motivation:

Major depressive disorder (MDD) affects twice as many women as men and women are at an increased risk during hormonal transition phases such as pregnancy and birth. A highly relevant subpopulation within the mixed MDD diagnostic category comprises women who develop perinatal depression (PND). PND is defined as a depressive episode with onset during pregnancy or up to 4 weeks postpartum, however epidemiological studies show that the risk of developing depression is heightened for 6 months postpartum. PND affects 10-15% of mothers postpartum. Why certain women are at high risk of developing perinatal depression (PND) remains unclear but recent studies suggest that these women might be particularly sensitive to the transition from high levels of placenta-produced sex-steroids in pregnancy to the hormone withdrawal phase postpartum. Further, pharmacologically induced changes in ovarian sex-hormones can produce depressive symptoms in a subgroup of otherwise healthy women and that the emergence of depressive symptoms is linked to both estrogen fluctuations and increases in serotonin transporter (SERT) brain binding (which putatively lowers serotonergic brain tone). Intriguingly, common gene variants that index SERT expression levels show "gene BY environment" associations with risk for depression, such that high-expressing SERT genotypes render women more vulnerable to depressive symptoms early - but not late - postpartum in a "gene-dose" dependent manner. Further, DNA methylation and gene expression markers of estradiol sensitivity predispose to PND and are linked to the estradiol stimulation phase in the pharmacological manipulation of sex-steroids risk model, thus constituting a candidate biomarker for PND.

It is currently unknown if estradiol sensitivity during pregnancy confers to PND risk through mechanism that (transiently) affect serotonergic tone in susceptible women. Changes in brain function late in pregnancy may extend to the early postpartum and shape how the brain integrates additional neurobiological changes that are associated with the postpartum hormonal withdrawal phase. This study will examine these mechanisms in a group of pregnant women that are followed from late pregnancy across early to late postpartum up to 6 month.

Natural variation in SERT-genotypes provides a unique opportunity to specifically address the interaction between SERT-gene expression-capacity and estradiol exposure through pregnancy in processes driving changes in serotonergic tone, brain structure and activity, and mental health from late pregnancy to 6 months postpartum. The time-points comprise: basic program: 2-5 days postpartum, 6 weeks postpartum and 6 months postpartum for all participants and for the imaging program participants: 2-5 days postpartum, 3-5 weeks postpartum, 12 weeks postpartum, 6 months postpartum.

By including women who undergo planned caesarean section, cerebrospinal fluid (CSF) can be obtained and thus, for the first time combine CSF markers of serotonergic tone and other transmitter systems (serotonin, 5-hydroxyindolacetic acid, other monoamines, γ-aminobutyric acid) with molecular brain imaging methods that index serotonergic tone (i.e. serotonin 4 receptor binding)

Aims:

* Determine if depressive symptoms from late pregnancy to 6 months postpartum map onto molecular brain imaging markers of serotonin signaling early postpartum (week 3-5), and evaluate if such markers and/or symptoms are dependent on serotonin transporter genotype and/or predicted by candidate gene transcription biomarkers for estrogen sensitivity.
* Evaluate how markers of stress-regulation capacity, brain activity, brain structure (hippocampal volume) and central markers of neurotransmission are associated with the emergence of depressive symptoms in women postpartum.
* Map the association between serotonin-4 receptor binding and cerebrospinal fluid markers of serotonergic tone (serotonin and 5-hydroxyindolacetic acid levels).
* Determine if markers of mental distress in women during pregnancy and the postpartum period are associated with infant markers of stress-regulation and serotonergic signaling in placenta and umbilical cord blood.

Hypotheses:

* Women with high-expressing SERT genotypes are more sensitive to estradiol exposure in late pregnancy in terms of changes in proxies for serotonergic tone (PET imaging or csf based) and emergence of depressive symptoms in late pregnancy and/or postpartum and such an association will be stronger in the presence of candidate gene transcript PND biomarkers.
* CSF levels of 5-hydroxyindolacetic acid are associated with serotonin 4 receptor brain PET (Positron Emission Tomography) binding.

Study design:

150 pregnant women between 18-40 years of age who deliver by planned caesarean section, due to breech presentation of the fetus or previous caesarean section, will be included in a longitudinal study. Participants will be recruited at the midwife clinic of Rigshospitalet, Copenhagen, Denmark. Based on natural variation in European populations the expected distribution of high vs. low expressing SERT genotypes is 40/60, respectively, thus genotype status can be included in the analysis structure. Self-reported psychometrics and questionnaires will be collected online at inclusion, across the pre- to postpartum transition and up to 6 months postpartum (basic program: 2-5 days postpartum, 6 weeks postpartum and 6 months postpartum; imaging program: 2-5 days postpartum, 3-5 weeks postpartum, 12 weeks postpartum, 6 months postpartum). CSF will be collected as part of the anesthetic procedures for a planned caesarean section, thus avoiding any additional invasive procedures. CSF markers of serotonergic tone (serotonin and its main metabolite, 5-HIAA) will be measured by HPLC techniques. Corresponding blood samples for determining relevant biomarkers (sex-steroids, DNA, mRNA and microRNA) and saliva for hypothalamic-pituitary-adrenal axis dynamics, will be taken just before the planned caesarean section. Hair from mother and infant will be collected around delivery for further cortisol analyses. Placenta tissue and umbilical cord blood will also be collected for determining relevant markers of serotonergic and hypothalamic-pituitary-adrenal axis functioning.

A subgroup of the study cohort selected towards high (N=35) or low risk for later manifest PND (N=35), based on symptoms of mental distress 2-5 days postpartum (in-house interview, high-risk scores correspond to at least 12 on the Kennerley Maternity Blues Questionnaire and at least 8 on Stein's Maternity Blues Scale), will participate in an extended brain imaging program. This program will include 5-HT4R ([11C]SB207145) PET, structural MRI, functional MRI (including emotional processing, reward processing and resting state fMRI), neuropsychological testing and face to face rating of mental state with a semi-structured interview (HAM-D17).

The study includes long-term follow-up at six months. Collected data will enter the Center for Integrated Molecular Brain Imaging database, thus providing a basis for longitudinal follow-up, data sharing and crossvalidation.

Statistics:

Power calculations based on inter-subject variability of the 5-HT4R show that an imaging group size of 35 is required to detect a 15% difference with a power of 0.8 for the brain regions of interest. With the full cohort number of 150 and due to oversampling of high and low risk women, about 25 women are expected to develop manifest PND episodes and more will display subclinical depressive symptoms, which will allow for correlation analyses with relevant outcome parameters including the candidate gene transcript based biomarker of estrogen sensitivity.

Highly correlated self-reported psychometric outcomes will be included in a latent variable construct of self-reported mental state (composite measure) using structural equation modelling.

Ethics:

The PET scans convey no known risk for adults. Infants will not be exposed to radiation and will be nursed by special staff or a close relative while the mother is scanned. Participants who develop levels of mental distress or depressive symptoms that approach clinical thresholds will be referred to relevant and timely psychiatric care. The study has been approved by the local ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Healthy pregnant women planned to deliver by caesarean section due to breech position of the fetus or previous caesarean section.

Exclusion Criteria:

* Current or previous severe psychiatric disorder such as psychotic disorders, eating disorder and bipolar disorder or current or previous psychiatric disorder requiring hospitalization.
* Current or previous neurological diseases, severe somatic disease, severe postpartum hemorrhage or use of medication that can interfere with study outcomes
* Severe disease or malformations in infants
* Obesity or underweight (pre-gestational BMI below 18 or above 35)
* Not fluent in Danish or severe visual or hearing impairments
* Earlier or present learning disabilities
* MRI contraindications (claustrophobia, metal implants)
* Previous exposure to radioactivity > 10 millisievert (mSv) within the last year
* Alcohol or drug abuse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the midwife clinic at Rigshospitalet, Copenhagen, i.e., included women will be residents of the central Copenhagen area.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Week 3-6 postpartum
  Edinburgh Postnatal Depression Scale. Score range: 0-30. Higher scores indicate more symptoms of postpartum depression. Total group
Depressive symptoms | Week 3-6 postpartum
  Score on the Hamilton 17-item depression scale. Score range: 0-52. Higher scores indicate more depressive symptoms. Assessed in imaging group
Gene transcript and DNA methylation markers of estrogen sensitivity | Prior to caesarean section
  116 a priori defined gene transcripts, which where differentially expressed in third trimester of women who later developed perinatal depression with postpartum onset relative to pregnant women who did not and to other depressed (reference Mehta et al, 2014, Psychological Medicine) and confirmed to be coupled to estrogen fluctuations (Mehtaet al. 2018 British Journal of Psychiatry) will be evaluated in the total group.
  Also DNA methylation of the genes of these transcripts will be determined and analysed in terms of their predictive value (above chance) for perinatal depression.
Cerebral serotonin 4 receptor binding postpartum | Week 3-6 postpartum
  Latent variable construct of brain 5-HT4R level based on quantification of 5-HT4R binding from 11C-SB207145 positron emission tomography in primary volumes of interest; neocortex, nucleus caudatus, putamen and hippocampus. Assessed in imaging group.
CSF levels of GABA | On day of caesarean section
  Assessed in total group
CSF levels of serotonin metabolite (5-HIAA) | On day of caesarean section
  Assessed in total group
Cortisol awakening response | Week 3-6 postpartum
  Cortisol awakening response, area under the curve with respect to baseline from 0 to 60 minutes from awakening.
Hair cortisol level mothers | On day of caesarean section.
  Provides an estimate of cortisol exposure up to 6 months prior to delivery, total group
Hair cortisol level newborns | Day 0-5 postpartum.
  Provides an estimate of fetal cortisol exposure, infants from total group
Hippocampal volumes | Week 3-6 postpartum.
  Hippocampal brain volume (including hippocampus) from structural MRI, imaging group.
functional MRI response to reward | Week 3-6 postpartum.
  fMRI (BOLD response) based assessment of brain activity in response to reward, relative to non-reward, stimuli. Assessed in imaging cohort
Resting state functional connectivity MRI | Week 3-6 postpartum
  rsfMRI based spontaneous co-fluctuations in low frequency BOLD signal, (functional connectivity). Assessed with rsfMRI scan in the resting state, i.e. non-goal oriented spontaneous thought and awake. Assessed in imaging group.
Change in epigenetic SERT status | From just before delivery to 3-6 weeks postpartum
  Change in epigenetic SERT status from late pregnancy to postpartum week 3-6.
Concentration of inflammatory markers, i.e hsCRP and immunoactive cytokines, in peripheral blood | At week 3-6
  Composite measure of hsCRP, TNF-α, IL-6, IL-18 and IL-10 levels, total group
functional MRI response to emotional faces | Week 3-6 postpartum.
  fMRI (BOLD response) based assessment of brain activity to emotionally salient, relative to neutral, stimuli. Assessed in imaging cohort.

SECONDARY OUTCOMES:
Depressive symptoms | Day 3-5 postpartum
  Score on the Hamilton 17-item depression scale. Score range: 0-52. Higher scores indicate more depressive symptoms. Assessed in imaging group
Depressive symptoms | Week 12 postpartum
  Score on the Hamilton 17-item depression scale. Score range: 0-52. Higher scores indicate more depressive symptoms. Assessed in imaging group
Depressive symptoms | Day 3-5 postpartum
  Edinburgh Postnatal Depression Scale. Score range: 0-30. Higher scores indicate more symptoms of postpartum depression. Assessed in total group
Depressive symptoms | 6 months postpartum
  Edinburgh Postnatal Depression Scale. Score range: 0-30. Higher scores indicate more symptoms of postpartum depression. Assessed in all
CSF levels of serotonin | On day of caesarean section
  Assessed in total group
CSF levels of dopamine metabolites | On day of caesarean section
  Assessed in total group
CSF levels of noradrenaline metabolites | On day of caesarean section
  Assessed in total group
CSF levels of inflammatory markers | On day of caesarean section
  Composite measure of IFN-c, IFN-alfa TNF-alfa og IL-6, in total group
Estradiol level | Prior to caesarean section.
  Estradiol level in peripheral blood, total group
Estradiol level | At week 3-6 postpartum.
  Estradiol level peripheral blood, total group
Change in estradiol level | From baseline (caesarean section to week 3-6 postpartum)
  Estradiol change pre- to postpartum, peripheral blood total group
Progesterone level | Prior to caesarean section.
  Progesterone level in peripheral blood
Progesterone level | At week 3-6 postpartum.
  Progesterone level in peripheral blood
Change in progesterone level | From baseline (caesarean section to week 3-6 postpartum)
  Progesterone change pre- to postpartum, peripheral blood total group
Allopregnanolone level | Prior to caesarean section.
  Allopregnanolone level in peripheral blood
Allopregnanolone level | At week 3-6 postpartum.
  Allopregnanolone level in peripheral blood
Change in allopregnanolone level | From baseline (caesarean section to week 3-6 postpartum)
  Change in allopregnanolone level in peripheral blood
Change in cortisol level | From baseline (caesarean section to week 3-6 postpartum)
  Cortisol change pre- to postpartum, peripheral blood total group
Cortisol awakening response | Week 12 postpartum
  Cortisol awakening response, area under the curve with respect to baseline from 0 to 60 minutes from awakening.
Cortisol awakening response | Prior to caesarean section
  Cortisol awakening response, area under the curve with respect to baseline from 0 to 60 minutes from awakening.
Change in cortisol awakening response | ´From baseline (caesarean section to week 3-6 postpartum)
  Change in cortisol awakening response, from caesarean section to 3-6 weeks postpartum.
DNA methylation of the SERT gene | Prior to caesarean section
  Methylation status for the SERT gene, total group
DNA methylation of the SERT gene | Week 3-6 postpartum
  DNA Methylation status for the SERT gene, total group
DNA methylation of the FK506-binding protein 51 (FKBP5) gene | Prior to caesarean section.
  Methylation status for the FK506-binding protein 51 (FKBP5) gene, total group
DNA methylation of the FK506-binding protein 51 (FKBP5) gene | Week 3-6 postpartum
  Methylation status for the FK506-binding protein 51 (FKBP5) gene, total group
Change in DNA methylation of the FK506-binding protein 51 (FKBP5) gene | From baseline (caesarean section to week 3-6 postpartum)
  Change in methylation status for the FK506-binding protein 51 (FKBP5) gene from late pregnancy to postpartum week 3-6.
DNA methylation of the glucocorticoid receptor gene | Prior to caesarean section.
  Methylation status for the glucocorticoid receptor gene, total group
DNA methylation of the glucocorticoid receptor gene | Week 3-6 postpartum
  Methylation status for the glucocorticoid receptor gene, total group
Change in DNA methylation of the glucocorticoid receptor gene | From baseline (caesarean section to week 3-6 postpartum)
  Change in methylation status for the glucocorticoid receptor gene from late pregnancy to postpartum week 3-6.
DNA methylation of the COMT gene | Prior to caesarean section.
  Methylation status for the COMT gene, total group
DNA methylation of the COMT gene | Week 3-6 postpartum
  Methylation status for the COMT gene, total group
Change in DNA methylation of the COMT gene | From baseline (caesarean section to week 3-6 postpartum)
  Change in methylation status for the COMT gene from just before delivery to 3-6 weeks postpartum
DNA methylation of the MAO-A gene | Prior to caesarean section.
  Methylation status for the MAO-A gene, total group
Change in DNA methylation of the MAO-A gene | From baseline (caesarean section to week 3-6 postpartum)
  Change in methylation status for the MAO-A gene, total group
DNA methylation of the MAO-A gene | Week 3-6 postpartum
  Methylation status for the MAO-A gene, total group
DNA methylation of the oxytocin receptor gene | Prior to caesarean section.
  Methylation status for the oxytocin receptor gene, total group
DNA methylation of the oxytocin receptor gene | Week 3-6 postpartum
  Methylation status for the oxytocin receptor gene, total group
Change in DNA methylation of the oxytocin receptor gene | From baseline (caesarean section to week 3-6 postpartum)
  Change in methylation status for the oxytocin receptor gene, total group
DNA methylation of the oxytocin gene | Prior to caesarean section.
  Methylation status for the oxytocin gene, total group
DNA methylation of the oxytocin gene | Week 3-6 postpartum
  Methylation status for the oxytocin gene, total group
Change in DNA methylation of the oxytocin gene | From baseline (caesarean section to week 3-6 postpartum)
  Change methylation status for the oxytocin gene, total group
Systemic inflammation peripheral blood hsCRP and immunoactive cytokines | Prior to caesarean section.
  Composite measure of hsCRP, TNF-α, IL-6, IL-18 and IL-10 levels, total group
Change in systemic inflammation peripheral blood hsCRP and immunoactive cytokines | From baseline (caesarean section to week 3-6 postpartum
  Change in composite measure of hsCRP, TNF-α, IL-6, IL-18 and IL-10 levels, total group
Self reported family history of mood disorders | Day 3-5 postpartum or before
  Family History Assessment Module (OS-FHAM). Number of first degree relatives with a history of depressive episodes or bipolar disorder. Total group.
Self reported impulsiveness score | Day 3-5 postpartum or before
  Barratt Impulsiveness Scale (BIS-11), self-reported. Range: 30-120. Total group.
Self reported Neuroticism score from NEO personality questionnaire | Day 3-5 postpartum or before
  NEO-PI-R - Revised NEO Personality Inventory, self-reported. Participants may score 20-80 for each of the personality traits: openness, conscientiousness, extraversion, agreeableness, and neuroticism. The higher the score, the more prominent is the personality trait. Total group.
Self reported parental bonding quality | Day 3-5 postpartum or before
  Parental bonding instrument (PBI), both parents, self-reported. Total group.
Self-reported perceived stress | Day 3-5 postpartum
  Perceived Stress Scale (PSS), range 0-40, a score of 0 indicates no perceived stress. Total group.
Self-reported perceived stress | Week 3-6 postpartum
  Perceived Stress Scale (PSS), range 0-40, a score of 0 indicates no perceived stress. Total group.
Change in self-reported perceived stress | Change from day 3-5 to week 3-6 postpartum
  Change in Perceived Stress Scale (PSS), range 0-40, a score of 0 indicates no perceived stress. Total group.
Self-reported anhedonia | Day 3-5 postpartum
  Snaith-Hamilton Pleasure Scale (SHAPS), range 0-14, a score of 0 indicates no self-reported anhedonia. Total group.
Self-reported anhedonia | Week 3-6 postpartum
  Snaith-Hamilton Pleasure Scale (SHAPS), range 0-14, a score of 0 indicates no self-reported anhedonia. Total group.
Change in self-reported anhedonia | Change from day 3-5 to week 3-6 postpartum
  Change in Snaith-Hamilton Pleasure Scale (SHAPS) score, range 0-14, a score of 0 indicates no self-reported anhedonia. Total group.
Self-reported rumination | Day 3-5 postpartum
  Rumination Response Scale (RRS), range 22-88, a score of 22 indicates no ruminative symptoms. Total group.
Self-reported rumination | Week 3-6 postpartum
  Rumination Response Scale (RRS), range 22-88, a score of 22 indicates no ruminative symptoms. Total group.
Change in elf-reported rumination | Change from day 3-5 to week 3-6 postpartum
  Change in Rumination Response Scale (RRS) score, range 22-88, a score of 22 indicates no ruminative symptoms. Total group.
Self-reported mood | Day 3-5 postpartum
  Profile of Mood States (POMS), range 0-260, a score of 0 indicates no mood disturbance. Total group.
Self-reported mood | Week 3-6 postpartum
  Profile of Mood States (POMS), range 0-260, a score of 0 indicates no mood disturbance. Total group.
Change in self-reported mood | Change from day 3-5 to week 3-6 postpartum
  Change in Profile of Mood States (POMS) score, range 0-260, a score of 0 indicates no mood disturbance. Total group.
Self-reported sleep quality | Day 3-5 postpartum
  Pittsburgh Sleep Quality Index (PSQI), range 0-21, a score of 0 indicates a healthy sleep quality. Total group.
Self-reported sleep quality | Week 3-6 postpartum
  Pittsburgh Sleep Quality Index (PSQI), range 0-21, a score of 0 indicates a healthy sleep quality. Total group.
Change in self-reported sleep quality | Change from day 3-5 to week 3-6 postpartum
  Change in Pittsburgh Sleep Quality Index (PSQI), range 0-21, a score of 0 indicates a healthy sleep quality. Total group.
Self-reported psychiatric symptoms | Day 3-5 postpartum
  Brief symptom Inventory-53 item (BSI-53), range 0-212, increasing score means worsening of symptoms.Total group.
Self-reported psychiatric symptoms | Week 3-6 postpartum
  Brief symptom Inventory-53 item (BSI-53), range 0-212, increasing score means worsening of symptoms.Total group.
Change in self-reported psychiatric symptoms | Change from day 3-5 to week 3-6 postpartum
  Change in Brief symptom Inventory-53 item (BSI-53) score, range 0-212, increasing score means worsening of symptoms.Total group.
Self-reported well-being | Day 3-5 postpartum
  WHO-5 well-being index, range 0-100, low score means less well-being. Total group.
Self-reported well-being | Week 3-6 postpartum
  WHO-5 well-being index, range 0-100, low score means less well-being. Total group.
Change in self-reported well-being | Change from day 3-5 to week 3-6 postpartum
  Change in WHO-5 well-being index, range 0-100, low score means less well-being. Total group.
Self-reported anxiety | Day 3-5 postpartum
  State Trait Anxiety Inventory (STAI-AD-D), state and trait subscales each have a range of 20-80, 20 means no anxiety. Total group.
Self-reported anxiety | Week 3-6 postpartum
  State Trait Anxiety Inventory (STAI-AD-D), state subscale range 20-80, 20 means no anxiety. Total group.
Change in self-reported anxiety | Change from day 3-5 to week 3-6 postpartum
  Change in State Trait Anxiety Inventory (STAI-AD-D) score, state subscale range 20-80, 20 means no anxiety. Total group.
Self-reported obsessive and compulsive symptoms | Day 3-5
  Obsessive-Compulsive Inventory (OCI) score, self-reported, range 0-72, higher scores indicate more symptoms. Total group.
Self-reported obsessive and compulsive symptoms | Week 3-6 postpartum
  Obsessive-Compulsive Inventory (OCI) score, self-reported, range 0-72, higher scores indicate more symptoms. Total group.
Change in self-reported obsessive and compulsive symptoms | Change from day 3-5 to week 3-6 postpartum
  Change in Obsessive-Compulsive Inventory (OCI) score, self-reported, range 0-72, higher scores indicate more symptoms. Total group.
Performance on Simple Reaction Time | Week 3-6 postpartum
  Performance on Simple Reaction Time, in imaging cohort.
Gray matter brain volume prefrontal cortex and anterior cingulate cortex | At week 3-6 postpartum
  Gray matter brain volume prefrontal cortex and anterior cingulate cortex
Serotonergic turnover in placenta | At delivery.
  Composite measure of serotonin, tryptophan og tryptofan hydroxylase levels relative to 5-HIAA, in placenta sample. Infants from total group
11-beta-hydroxysteroid dehydrogenase type 2 activity in placenta | At delivery
  11-beta-hydroxysteroid dehydrogenase type 2 activity in placenta. Infants from total group
Methylation status of genes relevant for stress-hormone regulation in placenta | At delivery
  Composite measure of methylation status for the FKBP5, glucocorticoid receptor, 11-beta hydroxysteroid dehydrogenase type 2 genes. Infants from total group
Methylation status of genes related to serotonergic signaling in placenta | At delivery
  Composite measure of the methylation status for monoamine oxidase, serotonin receptor and serotonin transporter genes. Infants from total group
Methylation status and gene transcript profiles of relevance for early brain development and stress regulation in newborn infants | At delivery.
  Composite measure of methylation status and gene transcript profiles of Glucocorticoid receptor, FKBP5, oxytocin and oxytocin receptors, Brain-derived neurotrophic factor (BDNF) genes. Assessed in blood from umbilical cord blood sample from infants, total group.

OTHER OUTCOMES:
COMT-genotype (rs4680) variant, i.e met/met vs other polymorphisms | Prior to caesarean section.
  val158met (rs4680) status, binary variable, i.e. "val/val, val/met" vs "met/met" variants
BDNF genotype (rs6265) status, i.e. val/val versus met-carrier variants | Prior to caesarean section.
  BDNF val66met (rs6265) status, binary variable, i.e. "val/val" versus "met-carrier" status
5-HTT genotype status, i.e LALA vs low-expressing (S or LG) variants | Prior to caesarean section.
  5-HTTLPR genotype status (binary), i.e. high-expressing LALA vs low-expressing (S or LG) variants, based on SLC6A4, i.e. L or S variants, and further subtyping on rs25531 haplotype L(A)L(A) vs LGLA, LGLG or variants containing as S as specified above.
Postpartum blues symptoms | Day 3-5 postpartum.
  In house interview based on Kennerley Maternity Blues Questionnaire, range: 0-28, higher score indicates more severe postpartum blues symptoms. High blues score is associated with greater risk for perinatal depression at week 3-6.
Postpartum blues symptoms | Day 3-5 postpartum.
  In house interview based on Stein's Maternity Blues Scale, range 0-26. High blues score is associated with greater risk for perinatal depression at week 3-6.

CONTACTS AND LOCATIONS:
Overall Officials: Vibe Frokjaer, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Via database of Center for Integrated Molecular Brain Imaging (Knudsen et al 2016, NeuroImage) data will be available for neuroscience research community contingent on approval by scientific board.
Supporting Information: Study Protocol
Time Frame: 2020-2035
Access Criteria: Approval by scientific board

REFERENCES:
- [Background] Carpenter LL, Anderson GM, Siniscalchi JM, Chappell PB, Price LH. Acute changes in cerebrospinal fluid 5-HIAA following oral paroxetine challenge in healthy humans. Neuropsychopharmacology. 2003 Feb;28(2):339-47. doi: 10.1038/sj.npp.1300025. PMID 12589387
- [Background] Caspi A, Hariri AR, Holmes A, Uher R, Moffitt TE. Genetic sensitivity to the environment: the case of the serotonin transporter gene and its implications for studying complex diseases and traits. Am J Psychiatry. 2010 May;167(5):509-27. doi: 10.1176/appi.ajp.2010.09101452. Epub 2010 Mar 15. PMID 20231323
- [Background] Guintivano J, Arad M, Gould TD, Payne JL, Kaminsky ZA. Antenatal prediction of postpartum depression with blood DNA methylation biomarkers. Mol Psychiatry. 2014 May;19(5):560-7. doi: 10.1038/mp.2013.62. Epub 2013 May 21. PMID 23689534
- [Background] Haahr ME, Fisher PM, Jensen CG, Frokjaer VG, Mahon BM, Madsen K, Baare WF, Lehel S, Norremolle A, Rabiner EA, Knudsen GM. Central 5-HT4 receptor binding as biomarker of serotonergic tonus in humans: a [11C]SB207145 PET study. Mol Psychiatry. 2014 Apr;19(4):427-32. doi: 10.1038/mp.2013.147. Epub 2013 Nov 5. PMID 24189342
- [Background] Klengel T, Binder EB. Gene-environment interactions in major depressive disorder. Can J Psychiatry. 2013 Feb;58(2):76-83. doi: 10.1177/070674371305800203. PMID 23442893
- [Background] Knudsen GM, Jensen PS, Erritzoe D, Baare WFC, Ettrup A, Fisher PM, Gillings N, Hansen HD, Hansen LK, Hasselbalch SG, Henningsson S, Herth MM, Holst KK, Iversen P, Kessing LV, Macoveanu J, Madsen KS, Mortensen EL, Nielsen FA, Paulson OB, Siebner HR, Stenbaek DS, Svarer C, Jernigan TL, Strother SC, Frokjaer VG. The Center for Integrated Molecular Brain Imaging (Cimbi) database. Neuroimage. 2016 Jan 1;124(Pt B):1213-1219. doi: 10.1016/j.neuroimage.2015.04.025. Epub 2015 Apr 17. PMID 25891375
- [Background] Marner L, Gillings N, Madsen K, Erritzoe D, Baare WF, Svarer C, Hasselbalch SG, Knudsen GM. Brain imaging of serotonin 4 receptors in humans with [11C]SB207145-PET. Neuroimage. 2010 Apr 15;50(3):855-61. doi: 10.1016/j.neuroimage.2010.01.054. Epub 2010 Jan 22. PMID 20096787
- [Background] Mehta D, Newport DJ, Frishman G, Kraus L, Rex-Haffner M, Ritchie JC, Lori A, Knight BT, Stagnaro E, Ruepp A, Stowe ZN, Binder EB. Early predictive biomarkers for postpartum depression point to a role for estrogen receptor signaling. Psychol Med. 2014 Aug;44(11):2309-22. doi: 10.1017/S0033291713003231. Epub 2014 Feb 5. PMID 24495551
- [Background] Mehta D, Rex-Haffner M, Sondergaard HB, Pinborg A, Binder EB, Frokjaer VG. Evidence for oestrogen sensitivity in perinatal depression: pharmacological sex hormone manipulation study. Br J Psychiatry. 2019 Sep;215(3):519-527. doi: 10.1192/bjp.2018.234. PMID 30457060
- [Background] Munk-Olsen T, Laursen TM, Pedersen CB, Mors O, Mortensen PB. New parents and mental disorders: a population-based register study. JAMA. 2006 Dec 6;296(21):2582-9. doi: 10.1001/jama.296.21.2582. PMID 17148723
- [Background] Sanjuan J, Martin-Santos R, Garcia-Esteve L, Carot JM, Guillamat R, Gutierrez-Zotes A, Gornemann I, Canellas F, Baca-Garcia E, Jover M, Navines R, Valles V, Vilella E, de Diego Y, Castro JA, Ivorra JL, Gelabert E, Guitart M, Labad A, Mayoral F, Roca M, Gratacos M, Costas J, van Os J, de Frutos R. Mood changes after delivery: role of the serotonin transporter gene. Br J Psychiatry. 2008 Nov;193(5):383-8. doi: 10.1192/bjp.bp.107.045427. PMID 18978318